CLINICAL TRIAL: NCT06901284
Title: Graded Exercise Hypoxia Testing
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael J. Joyner, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 25-000497
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 50 participants (25 female, 25 male) who are physically active for at least 150 minutes per week, at a moderate activity level.
  Interventions: Diagnostic Test: Graded Exercise Test; Diagnostic Test: Graded Hypoxia Exercise Test

INTERVENTIONS:
Diagnostic Test: Graded Exercise Test — Participants will perform a graded exercise test on either a cycle ergometer or treadmill. The testing protocol will begin with a 5- 10 min warm-up of either cycling or running/walking at the participants preferred pace.
  If the graded exercise test is on a bike, exercise will begin at wattage that elicits ~50% of their heart rate max, HRmax = 208 - 0.7 × age and increase by either 10W, 15W, or 20W every two minutes in a stepwise fashion until symptom limitation. The step of the wattage increase will be at the discretion of the investigators.
  If the graded exercise test is on a treadmill, the test will begin at a speed that elicits ~50% of predicted HRmax. Following, the speed of the treadmill will increase 0.5 mph (0.8 km/hr) every two minutes in a stepwise fashion until symptom limitation. If the participant maxes out the speed of the treadmill, we will increase the grade 2% every 2-minutes until symptom limitation.
Diagnostic Test: Graded Hypoxia Exercise Test — Participants will perform a single constant work rate exercise tests during graded hypoxia. They will be outfitted with either a facemask or mouthpiece connected to a uni-directional breathing valve. During inspiration, subjects will breathe from a closed-system Douglas bag balloon reservoir (~200 L) connected to the value on the inspired side via air-tight clean-bor tubing.
  The participant will complete the same mode of exercise as they did during visit 1, either bike or treadmill. The resistance on the bike or incline of the treadmill will be set to elicit an intensity equivalent to ~50% of their V̇O2max determined during visit 1. Participants will complete 5-minute stages over a range of FiO2 values. The exercise test will begin in an FiO2=0.21 (i.e. room air). Following this first 5-min stage the FiO2 will increase to 0.25, afterwards, participants will complete another stage at FiO2=0.21 and then decrease in a stepwise fashion every 5-minutes.

SUMMARY:
The purpose of this study is to develop a single, standardized test to determine how individuals tolerate acute hypoxia in a stepwise fashion. We aim to evaluate the association between multiple factors, such as ventilatory compensation, heart rate response, acid-base changes, sex, pulmonary function, etc, which may explain why some individuals tolerate exercise in hypoxia better than others. Identifying these factors of association will inform future pharmacological and non-pharmacological attempts to combat acute hypoxic exercise.

ELIGIBILITY:
Inclusion Criteria:

• Physically active (≥150 minutes of moderate physical activity per week)

Exclusion Criteria:

* Contraindications to exercise testing
* Currently pregnant
* Musculoskeletal or metabolic disease
* Allergies to lidocaine
* Body-mass index ≤18 or ≥35 kg·m-2
* Pacemaker
* No confounding cardiorespiratory disease
* Persistent tobacco use (>15 pack years)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 50 participants (25 female, 25 male) will be recruited for this study. Participants will be recruited from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04-24 (Estimated); Study Completion 2028-04-24 (Estimated)

PRIMARY OUTCOMES:
PaO₂/FiO₂ Ratio | 30 minutes
  The PaO₂/FiO₂ ratio is a widely used measure of oxygenation efficiency in the lungs. It compares the arterial oxygen partial pressure (PaO₂, measured in mmHg) to the fraction of inspired oxygen (FiO₂, expressed as a decimal). The ratio provides insight into the ability of the lungs to transfer oxygen into the bloodstream. A PaO₂/FiO₂ ratio of 300-400 is considered to be mild hypoxemia. Participants are considered as poorly tolerating hypoxia if their ratio is <400 and good at tolerating hypoxia if their ratio is >400.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Joyner, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - St. Mary's Hospital, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No